CLINICAL TRIAL: NCT02047110
Title: A 48 Weeks, Phase II, Randomized, Double-blind, Placebo-controlled, Proof of Concept and Dose Finding Study of Three Different Dose Regimens of BI 655066 Administered Subcutaneously in Patients With Ankylosing Spondylitis.
Brief Title: BI 655066 (Risankizumab) Proof of Concept Dose Finding Study in Ankylosing Spondylitis (AS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1311.8; 2013-003666-13 (EudraCT Number)
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Ankylosing Spondylitis (AS)
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — risankizumab

ARMS (4):
- Placebo (Placebo Comparator): Subcutaneous injection of Placebo (solution for injection matching risankizumab, 1 mL pre-filled syringe) administered every 8 weeks (At Day1 and at Weeks 8, 16, and 24) up to 4 times during the regular treatment period.
  Interventions: Drug: placebo for risankizumab
- Risankizumab 18 mg (Experimental): Subcutaneous injection of risankizumab 18 mg administered every 8 weeks at Day 1 only, followed by placebo every 8 weeks (i.e. at Week 8, 16 and 24), up to a total duration of 24 weeks
  Interventions: Drug: risankizumab
- Risankizumab 90 mg (Experimental): Subcutaneous injection of risankizumab 90 mg administered every 8 weeks (At Day1 and at Weeks 8, 16, and 24) up to 4 times during the regular treatment period
  Interventions: Drug: risankizumab
- Risankizumab 180 mg (Experimental): Subcutaneous injection of risankizumab 180 mg administered every 8 weeks (At Day1 and at Weeks 8, 16, and 24) up to 4 times during the regular treatment period
  Interventions: Drug: risankizumab

INTERVENTIONS:
Drug: placebo for risankizumab — Placebo for risankizumab administered by subcutaneous (SC) injection
  Arms: Placebo
Drug: risankizumab — Risankizumab administered by subcutaneous (SC) injection
  Other Names: ABBV-066; BI 655066; SKYRIZI
  Arms: Risankizumab 18 mg; Risankizumab 180 mg; Risankizumab 90 mg

SUMMARY:
The overall purpose of the trial is to assess the clinical efficacy of three different subcutaneous doses of BI 655066 (risankizumab) in adult patients with AS, in order to provide clinical proof of concept and to select dose (s) for confirmatory clinical trials.

ELIGIBILITY:
Inclusion criteria:

1. Male and female patients
2. Age = 18 years and = 70 years
3. Definite AS based on the modified New York criteria (1984)
4. Documented disease duration = 3 months at screening
5. Active disease at screening, defined as:

   1. BASDAI score (0-10) = 4, AND
   2. Spinal pain level assessed by the 2nd BASDAI question (0-10) = 4
6. Have either a documented inadequate response for axial symptoms to 30 days of optimal daily doses of at least two non-steroidal anti-inflammatory drugs (NSAIDs), or documented intolerance to NSAIDs
7. Female patients who meet any of the following criteria from screening visit up to the End of Observation visit (EOO):

   * using adequate contraception, e.g. any of the following methods plus condom: implants, injectables, combined oral contraceptives, intrauterine device (IUD)
   * sexually abstinent
   * have a vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
   * surgically sterilised (including hysterectomy)
   * postmenopausal defined as at least 1 year of spontaneous Amenorrhea
8. Patients (males or females) receiving background MTX or Leflunomide therapy who are following the national regulatory guidelines regarding contraception
9. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion criteria:

1. Radiographic evidence of total ankylosis of the spine at screening or before (spinal XRay examinations at screening visit/ during screening period are not mandatory ¿ see footnote 12 from Flow-Chart 1)
2. Patient previously treated with any biological immunomodulating agent for AS, either licensed or experimental
3. Previous or current participation in a clinical trial testing an investigational drug for AS within 12 weeks prior to randomization (any biological immunomodulating agents are excluded)
4. Usage of any investigational drug within 30 days prior to randomization or the planned use of an investigational drug during the course of the actual study
5. Active uveitis or inflammatory bowel disease at screening
6. Diagnosed psoriatic arthritis at screening, satisfying the modified New York criteria
7. Patients who had received intraarticular injection(s) with corticosteroids within 4 weeks prior to screening visit
8. Patients who must or wish to continue the intake of restricted medications (cf. Section 4.2.2.1) or any drug considered likely to interfere with the safe conduct of the study
9. Major surgery performed within 8 weeks prior to screening or planned within 12 months after screening (e.g. hip replacement)
10. Chronic or relevant acute infections including HIV, viral hepatitis and tuberculosis (positive tests for HIV, HBV/HCV at screening will be exclusionary)

    For tuberculosis patients, they are not eligible according to the following screening criteria:
    * Have signs or symptoms suggestive of current active or latent TB upon medical history, physical examination and/or a chest radiograph (both posterior-anterior and lateral views, taken within 3 months prior to the first administration of study drug and read by a qualified radiologist)
    * Have history of latent or active TB prior to screening, except for patients who have documentation of having completed an adequate treatment regimen at least 6 months prior to the first administration of study agent
    * Have positive QuantiFERON-TB Gold In-Tube test within 2 months prior to or during screening, in which active TB has not been ruled out, except for patients with history of latent TB and documentation of having completed an adequate treatment regimen at least 6 months prior to the first administration of study agent
11. Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix
12. Evidence of current or previous clinically significant disease, medical condition other than AS, finding of the medical examination (including vital signs and ECG), or laboratory value at the screening visit outside the reference range that is of clinical relevance, that in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data. This criterion provides an opportunity for the investigator to exclude patients based on clinical judgment, even if other eligibility criteria are satisfied.
13. History of allergy/hypersensitivity to a systemically administered biologic agent or its excipients
14. History of alcohol abuse within last 12 months (intake of more than 30 g/day)
15. History of drug abuse within last 12 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2015-03-05 (Actual); Study Completion 2016-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

REFERENCES:
- [Derived] Baeten D, Ostergaard M, Wei JC, Sieper J, Jarvinen P, Tam LS, Salvarani C, Kim TH, Solinger A, Datsenko Y, Pamulapati C, Visvanathan S, Hall DB, Aslanyan S, Scholl P, Padula SJ. Risankizumab, an IL-23 inhibitor, for ankylosing spondylitis: results of a randomised, double-blind, placebo-controlled, proof-of-concept, dose-finding phase 2 study. Ann Rheum Dis. 2018 Sep;77(9):1295-1302. doi: 10.1136/annrheumdis-2018-213328. Epub 2018 Jun 26. PMID 29945918
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial had a double blind (DB) treatment period up to Week 24, an Escape treatment period up to Week 40, and an open-label-extension (OLE) treatment period that lasted 26 weeks after OLE entry. Each of the treatment periods was followed by a 24- week post-treatment follow-up period.
Period: DB Treatment Period up to Week 24
Arm/Group | Placebo | Risankizumab 18 mg | Risankizumab 90 mg | Risankizumab 180 mg
Started | 40 (Started are the treated patients) | 40 (Started are the treated patients) | 39 (Started are the treated patients) | 40 (Started are the treated patients)
Completed | 35 | 38 | 36 | 38
Not Completed | 5 | 2 | 3 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Other than specified | 1 | 2 | 3 | 1
Period: DB (Week 12 up to Week 24)
Arm/Group | Placebo | Risankizumab 18 mg | Risankizumab 90 mg | Risankizumab 180 mg
Started | 9 (Patients who continued treatment in the DB treatment period up to Week 24) | 17 (Patients who continued treatment in the DB treatment period up to Week 24) | 13 (Patients who continued treatment in the DB treatment period up to Week 24) | 12 (Patients who continued treatment in the DB treatment period up to Week 24)
Completed | 9 | 15 | 12 | 12
Not Completed | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Other than specified | 0 | 1 | 1 | 0
Period: Escape Treatment Period
Arm/Group | Placebo | Risankizumab 18 mg | Risankizumab 90 mg | Risankizumab 180 mg
Started | 26 (Assessment in SpondyloArthritis international Society (ASAS) 20 nonresponders) | 21 (ASAS 20 nonresponders) | 23 (ASAS 20 nonresponders) | 26 (ASAS 20 nonresponders)
Completed | 23 | 15 | 20 | 24
Not Completed | 3 | 6 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 1
Not completed — Adverse Event | 1 | 2 | 2 | 0
Not completed — Other than specified | 1 | 2 | 0 | 1
Period: OLE Treatment Period
Arm/Group | Placebo | Risankizumab 18 mg | Risankizumab 90 mg | Risankizumab 180 mg
Started | 4 (Patients with loss of ASAS 20 response compared with baseline) | 8 (Patients with loss of ASAS 20 response compared with baseline) | 5 (Patients with loss of ASAS 20 response compared with baseline) | 9 (Patients with loss of ASAS 20 response compared with baseline)
Completed | 4 | 8 | 4 | 9
Not Completed | 0 | 0 | 1 | 0
Not completed — Other than specified | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All patients who received at least 1 dose of trial medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Risankizumab 18 mg | Risankizumab 90 mg | Risankizumab 180 mg | Total
Number analyzed (Participants) | 40 | 40 | 39 | 40 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (11.0) | 38.0 (11.1) | 39.5 (10.8) | 40.6 (11.9) | 38.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 9 | 10 | 46
  Male | 25 | 28 | 30 | 30 | 113

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Achieved Assessment of Spondyloarthritis International Society (ASAS) 40 Improvement Criteria at Week 12.
Description: ASAS 40 evaluations are based on the following 4 components (also called domains) that include patient' self-assessments on a numerical rating scale (NRS) from 0 to 10 with higher numbers representing a worse disease status:
  * Global AS disease activity
  * Inflammation based on the mean of Bath AS Disease Activity Index (BASDAI) questions addressing the level of morning stiffness and duration
  * Spinal pain based on the mean of 2 questions
  * Physical function based on the Bath AS Functional Index (BASFI) The ASAS 40 response is defined as an improvement in 3 of 4 components and no worsening in the remaining component; an improvement is defined as a reduction from baseline of ≥40% and an absolute reduction of ≥2 units in each of the 3 components.
Time Frame: Week 12
Population: Full Analysis set (FAS): FAS comprised of all randomised patients who received at least 1 dose of trial medication
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Risankizumab 18 mg | Risankizumab 90 mg | Risankizumab 180 mg
Number analyzed (Participants) | 40 | 40 | 39 | 40
Percentage of participants | 17.5 | 25.0 | 20.5 | 15.0
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 18 mg; To control the type I error rate, the primary endpoint was tested in a hierarchical fixed sequence approach. The proportion of patients achieving ASAS 40 response at Week 12 was pairwise compared in the following sequence: risankizumab 180 mg vs. placebo (1.) and risankizumab 90 mg vs. placebo (2.). The significance level was 5% (1-sided). The comparison risankizumab 18 mg vs. placebo was not included in the formal testing sequence; an exploratory p-value was provided; Test type: Superiority or Other; p = 0.2652, Suissa-Shuster unconditional exact test — The Suissa-Shuster unconditional exact test was used to test the difference in the proportion of patients achieving the primary endpoint, ASAS 40 response at Week 12, between treatment groups; Risk Difference (RD) = 7.5, 90% CI 2-sided [-12.1 to 26.6] — The confidence interval for the difference in proportion between the treatment groups was obtained by the Clopper-Pearson method. Difference calculated as "risankizumab 18 mg minus Placebo"
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 90 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4129, Suissa-Shuster unconditional exact test — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 3.0, 90% CI 2-sided [-15.9 to 20.8] — The confidence interval for the difference in proportion between the treatment groups was obtained by the Clopper- Pearson method. Difference calculated as "risankizumab 90 mg minus Placebo"
Statistical Analysis 3: Comparison: Placebo vs Risankizumab 180 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4243, Suissa-Shuster unconditional exact test — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = -2.5, 90% CI 2-sided [-21.8 to 17.0] — The confidence interval for the difference in proportion between the treatment groups was obtained by the Clopper- Pearson method. Difference calculated as "risankizumab 180 mg minus Placebo"

2. Secondary Outcome: Change From Baseline to Week 12 in Disease Activity Assessed by the Ankylosing Spondylitis Disease Activity Score (ASDAS).
Description: This is the key secondary endpoint. ASDAS is a linear function of Back Pain (Question 2 from Bath Ankylosing Spondylitis (AS) Disease Activity Index (BASDAI): range 0-10), Duration of Morning Stiffness (Question 6 from BASDAI: range 0-10), Patient's global assessment of the disease on Numerical rating Scale (NRS) (range 0-10), peripheral joint pain/swelling (Question 3 from BASDAI: range 0-10) and the C-reactive protein (CRP) lab value at the visit. ASDAS-CRP: 0.121*Back pain +0.058*Duration of Morning Stiffness +0.11*Patient Global + 0.073*Peripheral pain/ Swelling + 0.579*Ln (CRP +1). For all of the scales that make up the ASDAS, higher indicates worse disease.
Time Frame: Baseline and Week 12
Population: FAS
Measure: Median (Inter-Quartile Range); unit: Unit on scale
Arm/Group | Placebo | Risankizumab 18 mg | Risankizumab 90 mg | Risankizumab 180 mg
Number analyzed (Participants) | 40 | 40 | 39 | 40
Unit on scale | -0.2 [-0.9 to 0.2] | -0.7 [-1.3 to -0.2] | -0.6 [-1.0 to 0.1] | -0.7 [-1.1 to -0.3]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 18 mg; Test type: Superiority or Other; p = 0.0229, Wilcoxon rank-sum test — One sided p-value from Wilcoxon rank-sum test; Median estimate by Hodges-Lehmann method = -0.4, 90% CI 2-sided [-0.7 to -0.1] — The confidence interval for the difference in proportion between the treatment groups was obtained by the Moses method. Difference calculated as "risankizumab 18 mg minus Placebo"
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 90 mg; Test type: Superiority or Other; p = 0.1038, Wilcoxon rank-sum test — One sided p-value from Wilcoxon rank-sum test; Median estimate by Hodges-Lehmann method = -0.3, 90% CI 2-sided [-0.6 to 0.1] — The confidence interval for the difference in proportion between the treatment groups was obtained by the Moses method. Difference calculated as "risankizumab 90 mg minus Placebo"
Statistical Analysis 3: Comparison: Placebo vs Risankizumab 180 mg; Test type: Superiority or Other; p = 0.0101, Wilcoxon rank-sum test — One sided p-value from Wilcoxon rank-sum test; Median estimate by Hodges-Lehmann method = -0.5, 90% CI 2-sided [-0.7 to -0.1] — The confidence interval for the difference in proportion between the treatment groups was obtained by the Moses method. Difference calculated as "risankizumab 180 mg minus Placebo"

3. Secondary Outcome: Percentage of Patients Who Achieved ASAS 5/6 Improvement Criteria at Week 12
Description: The ASAS 5/6 evaluation is based on 6 components:
  * Global AS disease activity
  * Inflammation based on the mean of BASDAI questions addressing the level-of morning stiffness and duration
  * Spinal pain
  * Physical function based on the Bath AS Functional Index (BASFI)
  * Spinal mobility assessment (lateral lumbar flexion), corresponding to one out of 5 measurements of Bath Ankylosing Spondylitis Metrology Index (BASMI)
  * Serum CRP levels The ASAS 5/6 response is defined as an improvement in any 5 of the 6 components and no worsening in the remaining component. A reduction from baseline of ≥20% is defined as an improvement according to the ASAS criteria.
Time Frame: Week 12
Population: Full Analysis set (FAS): FAS comprised of all randomised patients who received at least 1 dose of trial medication
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Risankizumab 18 mg | Risankizumab 90 mg | Risankizumab 180 mg
Number analyzed (Participants) | 40 | 40 | 39 | 40
Percentage of participants | 5.0 | 20.0 | 23.1 | 17.5
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 18 mg; Test type: Superiority or Other; p = 0.0238, Suissa-Shuster unconditional exact test — The Suissa-Shuster unconditional exact test was used to test the difference in the proportion of patients achieving the endpoint at Week 12, between treatment groups; Risk Difference (RD) = 15.0, 90% CI 2-sided [-4.6 to 33.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 90 mg; Test type: Superiority or Other; p = 0.0120, Suissa-Shuster unconditional exact test — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 18.1, 90% CI 2-sided [-0.8 to 35.3] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs Risankizumab 180 mg; Test type: Superiority or Other; p = 0.0465, Suissa-Shuster unconditional exact test — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 12.5, 90% CI 2-sided [-7.1 to 31.4] — [estimate comment as in outcome 1, analysis 3]

4. Secondary Outcome: Percentage of Patients Who Achieved Partial Remission According to the ASAS Criteria at Week 12
Description: Percentage of patients who achieved partial remission according to the ASAS criteria at Week 12 is presented
Time Frame: Week 12
Population: Full Analysis set (FAS): FAS comprised of all randomised patients who received at least 1 dose of trial medication
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Risankizumab 18 mg | Risankizumab 90 mg | Risankizumab 180 mg
Number analyzed (Participants) | 40 | 40 | 39 | 40
Percentage of participants | 2.5 | 2.5 | 2.6 | 10.0
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 18 mg; p-values are not presented as they were not meaningful; 3 treatment groups had only a single patient with partial remission; Test type: Superiority or Other; Risk Difference (RD) = 0, 90% CI 2-sided [-19.4 to 19.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 90 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Risk Difference (RD) = 0.1, 90% CI 2-sided [-18.3 to 18.3] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs Risankizumab 180 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Risk Difference (RD) = 7.5, 90% CI 2-sided [-12.1 to 26.6] — [estimate comment as in outcome 1, analysis 3]

5. Secondary Outcome: Percentage of Patients Who Achieved ASAS 20 Improvement Criteria at Week 12
Description: ASAS 20 evaluations are based on the following 4 components (also called domains) that include patient' self-assessments on a numerical rating scale (NRS) from 0 to 10 with higher numbers representing a worse disease status:
  * Global AS disease activity
  * Inflammation based on the mean of Bath AS Disease Activity Index (BASDAI) questions addressing the level of morning stiffness and duration
  * Spinal pain based on the mean of 2 questions
  * Physical function based on the Bath AS Functional Index (BASFI) The ASAS 20 response is defined as an improvement in 3 of 4 components and no worsening in the remaining component; an improvement is defined as a reduction from baseline of ≥20% and an absolute reduction of ≥1 units in each of the 3 components.
Time Frame: Week 12
Population: Full Analysis set (FAS): FAS comprised of all randomised patients who received at least 1 dose of trial medication
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Risankizumab 18 mg | Risankizumab 90 mg | Risankizumab 180 mg
Number analyzed (Participants) | 40 | 40 | 39 | 40
Percentage of participants | 20.0 | 45.0 | 33.3 | 32.5
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 18 mg; Test type: Superiority or Other; p = 0.0092, Suissa-Shuster unconditional exact test — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 25.0, 90% CI 2-sided [5.5 to 43.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 90 mg; Test type: Superiority or Other; p = 0.1243, Suissa-Shuster unconditional exact test — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 13.3, 90% CI 2-sided [-5.9 to 30.5] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs Risankizumab 180 mg; Test type: Superiority or Other; p = 0.1198, Suissa-Shuster unconditional exact test — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 12.5, 90% CI 2-sided [-7.1 to 31.4] — [estimate comment as in outcome 1, analysis 3]

6. Secondary Outcome: Change From Baseline to Week 12 in Disease Activity Assessed by BASDAI
Description: BASDAI assesses the AS disease activity of a patient within the last week based on 6 questions on a NRS (1 to 10) How would you describe the overall level of
  1. fatigue/tiredness you have experienced?
  2. AS neck, back or hip pain you have had?
  3. pain/swelling in joints other than neck, back or hips you have had?
  4. discomfort you have had from any areas tender to touch or pressure?
  5. morning stiffness you have had from the time you wake up? How long does your
  6. morning stiffness last from the time you wake up?
  A score of 10 means very severe disease activity for each of the BASDAI questions 1, 2, 3, 4 and 5. BASDAI question 6 addresses the stiffness duration. A NRS of 0 means 0 h; a NRS of 10 mean ≥2 h.
  The BASDAI was computed in the following way: the sum of the values of question 1 to 4 was calculated and the mean of questions 5 and 6 was added. This value was divided by 5.
Time Frame: Baseline and Week 12
Population: FAS
Measure: Median (Inter-Quartile Range); unit: Unit on scale
Arm/Group | Placebo | Risankizumab 18 mg | Risankizumab 90 mg | Risankizumab 180 mg
Number analyzed (Participants) | 40 | 40 | 39 | 40
Unit on scale | -0.6 [-2.8 to -0.1] | -1.2 [-2.8 to -0.4] | -0.8 [-2.1 to 1.0] | -1.0 [-2.0 to -0.2]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 18 mg; Test type: Superiority or Other; p = 0.1241, Wilcoxon rank-sum test — One sided p-value from Wilcoxon rank-sum test; Median estimate by Hodges-Lehmann method = -0.4, 90% CI 2-sided [-1.0 to 0.2] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 90 mg; Test type: Superiority or Other; p = 0.3033, Wilcoxon rank-sum test — One sided p-value from Wilcoxon rank-sum test; Median estimate by Hodges-Lehmann method = 0.3, 90% CI 2-sided [-0.5 to 1.0] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs Risankizumab 180 mg; Test type: Superiority or Other; p = 0.3203, Wilcoxon rank-sum test — One sided p-value from Wilcoxon rank-sum test; Median estimate by Hodges-Lehmann method = -0.2, 90% CI 2-sided [-0.8 to 0.4] — [estimate comment as in outcome 2, analysis 3]

7. Secondary Outcome: Percentage of Patients Who Achieved ASAS 40 Improvement Criteria at Week 24
Description: Percentage of patients who achieved ASAS 40 improvement criteria at Week 24 is presented
Time Frame: Week 24
Population: Full Analysis set (FAS): FAS comprised of all randomised patients who received at least 1 dose of trial medication
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Risankizumab 18 mg | Risankizumab 90 mg | Risankizumab 180 mg
Number analyzed (Participants) | 40 | 40 | 39 | 40
Percentage of participants | 15.0 | 22.5 | 23.1 | 12.5
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 18 mg; Test type: Superiority or Other; p = 0.2639, Suissa-Shuster unconditional exact test — The Suissa-Shuster unconditional exact test was used to test the difference in the proportion of patients achieving the endpoint at Week 24, between treatment groups; Risk Difference (RD) = 7.5, 90% CI 2-sided [-12.1 to 26.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 90 mg; Test type: Superiority or Other; p = 0.2691, Suissa-Shuster unconditional exact test — [p-value comment as in outcome 7, analysis 1]; Risk Difference (RD) = 8.1, 90% CI 2-sided [-10.9 to 25.7] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs Risankizumab 180 mg; Test type: Superiority or Other; p = 0.4174, Suissa-Shuster unconditional exact test — [p-value comment as in outcome 7, analysis 1]; Risk Difference (RD) = -2.5, 90% CI 2-sided [-21.8 to 17.0] — [estimate comment as in outcome 1, analysis 3]

ADVERSE EVENTS:
Time Frame: All adverse events reported during the DB, the Escape, and the OLE treatment period; up to 50 weeks
Groups:
- Escape Low: Patients who received risankizumab 180 mg in the Escape treatment period and who were randomized to either Placebo or risankizumab 18 mg at Day 1 of the DB treatment period
- Escape High: Patients who received risankizumab 180 mg in the Escape treatment period and who were randomized to either risankizumab 90 mg or risankizumab 180 mg at Day 1 of the DB treatment period
- Escape: Patients who received escape treatments of risankizumab 180 mg regardless of the initial randomization group
- Open Label Extension (OLE): Patients who received 180 mg risankizumab (administered subcutaneously) every 8 weeks in OLE treatment period
- Risankizumab High: Patients who received at least one risankizumab 90 mg or 180 mg treatment during the entire trial
- Risankizumab Total: Patients who received at least one risankizumab treatment at any dose level
- Total_all: All randomised patients
Arm/Group | Placebo | Risankizumab 18 mg | Risankizumab 90 mg | Risankizumab 180 mg | Escape Low | Escape High | Escape | Open Label Extension (OLE) | Risankizumab High | Risankizumab Total | Total_all
Serious Adverse Events (participants affected / at risk) | 2/40 | 0/40 | 2/39 | 2/40 | 1/47 | 2/48 | 3/95 | 1/26 | 9/138 | 9/149 | 10/159
Other Adverse Events (participants affected / at risk) | 21/40 | 21/40 | 22/39 | 22/40 | 10/47 | 17/48 | 27/95 | 11/26 | 85/138 | 91/149 | 99/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | Risankizumab 18 mg (N=40) | Risankizumab 90 mg (N=39) | Risankizumab 180 mg (N=40) | Escape Low (N=47) | Escape High (N=48) | Escape (N=95) | Open Label Extension (OLE) (N=26) | Risankizumab High (N=138) | Risankizumab Total (N=149) | Total_all (N=159)
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1
Incision site cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | Risankizumab 18 mg (N=40) | Risankizumab 90 mg (N=39) | Risankizumab 180 mg (N=40) | Escape Low (N=47) | Escape High (N=48) | Escape (N=95) | Open Label Extension (OLE) (N=26) | Risankizumab High (N=138) | Risankizumab Total (N=149) | Total_all (N=159)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 3 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 1 | 1 | 2 | 0 | 8 | 8 | 8
Fatigue (General disorders) | 2 | 2 | 1 | 4 | 1 | 1 | 2 | 0 | 9 | 11 | 11
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 3 | 1 | 1 | 2 | 0 | 8 | 8 | 8
Gastroenteritis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 4 | 5 | 6
Influenza (Infections and infestations) | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 2 | 6 | 7 | 8
Nasopharyngitis (Infections and infestations) | 4 | 7 | 7 | 5 | 5 | 5 | 10 | 2 | 30 | 32 | 33
Sinusitis (Infections and infestations) | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 5 | 5 | 5
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 2 | 1 | 1 | 2 | 2 | 8 | 8 | 8
Wound (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 0 | 3 | 3 | 0 | 5 | 6 | 6
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 3 | 3 | 3
Blood creatine phosphokinase increased (Investigations) | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 5 | 5 | 7
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 3 | 3 | 3
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 1 | 5 | 6 | 1 | 8 | 9 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 6 | 6 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2 | 2 | 2 | 1 | 3 | 0 | 10 | 12 | 12
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 3 | 3 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 4 | 4 | 4
Headache (Nervous system disorders) | 3 | 5 | 3 | 4 | 2 | 1 | 3 | 0 | 14 | 15 | 17
Renal colic (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 3 | 3 | 3
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 0 | 2 | 2 | 2 | 7 | 7 | 7

LIMITATIONS AND CAVEATS:
The hierarchical testing p-values are exploratory in nature, due to the study design, as the primary endpoint of study failed to meet the desired objective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.